CLINICAL TRIAL: NCT05564845
Title: Brain Structure and Neurocognitive Development in Sickle Cell Disease; a Longitudinal Cohort Study (BRICK Study)
Acronym: BRICK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dr. Marjon H. Cnossen MD PhD (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Sponsor-Investigator, Dr. Marjon H. Cnossen MD PhD, Principal Investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-25022-0004
Record Dates: First submitted 2022-09-21; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Brain Development Abnormality; Sickle Cell Disease
Keywords: brain development; Sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Neurologic Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biobanking will take place prospectively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe SCD genotypes: Children between 6 and 18 years of age of genotypes HbSS, HbSβº
  Interventions: Diagnostic Test: MR scan of the brain; Diagnostic Test: Blood work; Diagnostic Test: Neurological examination; Diagnostic Test: Neuropsychological assessment
- Not severe SCD genotypes: Children between 6 and 18 years of age of genotypes HbSβ+, and HbSC and more
  Interventions: Diagnostic Test: MR scan of the brain; Diagnostic Test: Blood work; Diagnostic Test: Neurological examination; Diagnostic Test: Neuropsychological assessment

INTERVENTIONS:
Diagnostic Test: MR scan of the brain — Subjects will undergo MRI of the head, blood sampling and neurological examination on the same day or spread over 2 days. On a separate day from blood sampling and undergoing an MRI scan, the neuropsychological assessment will take place. The interval between the MRI scan and the neuropsychological assessment will be a maximum of 2 months. These measurements will be performed a total of 3 times with an interval of 2 years.
Diagnostic Test: Blood work — Lab work for current lab values and biobanking
Diagnostic Test: Neurological examination — Classical neurological examination
Diagnostic Test: Neuropsychological assessment — Overview of standard neurocognitive assessment tools in BRICK study Children and adolescents (Young) Adults
  * Wechsler Intelligence Test for Children- Fifth edition (WISC-V) (6-16 YOA) Wechsler Adult Intelligence Scale- Fourth edition WAIS-IV (16-24 YOA)
  * A Developmental NEuroPSYchological Assessment, Second Edition (NEPSY-II)
    * Narrative memory
    * Word fluency
    * Route finding NEPSY-II
  * World Fluency
  * Additional Questionnaires (6-18 years):
    * Child Behavior Checklist (CBCL)
    * Teacher Report Form (TRF)
    * Youth Self Report (YSR)
    * Behavior Rating Inventory of Executive Function (BRIEF), parent- and teacher-report)
    * Conners-3® • Additional Questionnaires (18+ years):
    * Adult Self-Report (ASR) / Adult Behavior Checklist (ABCL) (in case of IQ<70)
    * Behavior Rating Inventory of Executive Function Adult version (BRIEF-A), self-report / informant-report (in case of IQ<70)
    * Conners' Adult ADHD Rating Scales (CAARS)
  Emma toolbox

SUMMARY:
Sickle cell disease (SCD) is an autosomal recessive red blood cell blood disorder. One especially vital organ affected in SCD is the brain. Individuals with SCD have an increased risk of both overt cerebral infarctions and silent infarctions. The latter are brain lesions without apparent neurological sequelae. Since cortical neurons in the brain lack the ability to regenerate, tissue damage accumulates throughout the already shortened lifespan of individuals with SCD, resulting in far-reaching consequences such as significant cognitive impairment. Currently, only hematological stem cell transplantation can halt the multiorgan tissue damage. However, the criteria to determine the timing of curative therapy do not center the brain, despite that subtle anomalies of this critical organ can have long-lasting consequences. Since it is not yet known whether brain tissue damage precedes, parallels, or lags behind non-brain tissue damage, it is critical to map these effects in youth with SCD. While importantly comparing images with a healthy reference population. Understanding how the brain is affected is critical for clinical decision making, such as timing of potentially curative interventions but also, to prevent long term irreversible brain damage in youth with SCD. In this study, a cohort of 84 SCD patients between the ages of 6 and 18 at baseline, will undergo MR imaging, neurological examination, neuropsychological assessment and blood sampling three times in total, with intervals of two years; results will be innovatively compared with children included in the Generation R population study (±8000 MRIs children and (young)adults) 6-20 years of age). Our hypothesis, based on the inability of the brain to generate new cortical neurons following cell death, is that brain function is impaired earlier than other organ systems and that there is an age-dependent limit in the brain's ability to remodel itself based on neuroplasticity.

DETAILED DESCRIPTION:
Objective: The primary objective is to evaluate longitudinal developmental changes in brain structure in patients aged 6-18 years with SCD. The secondary objective is to analyze the longitudinal relations between biomarkers, demographic characteristics, brain structure, neurocognitive functioning, behavioral functioning and developmental changes in brain structure.

Study Design: Longitudinal cohort study (BRICK) with a duration of 4 years. Study population: Children and adolescents with sickle cell disease (SCD) of all genotypes (e.g. HbSS, HbSβº, HbSβ+, and HbSC) aged 6 -18 years. This will be compared to a cohort of healthy children and adolescents from Generation R.

Primary study endpoint:

* Total white matter volume increase in children and adolescents with SCD Secondary study endpoints
* Neurocognitive functioning (intelligence, specific neurocognitive functions, network organization)
* Incidence of stroke
* Other forms complications due to SCD
* Amount of hospital admissions, day care admissions (adult care only), crises at home, contact moments with the sickle cell center, ER visits
* Biomarkers for anemia, hemolysis, inflammation and endothelial activation.
* Behavioral functioning Nature and extent of the burden and risk associated with participation, benefit and group relatedness: By creating an advanced model for structural neurological, neurocognitive functioning in SCD, we will gain more insight into the pathophysiological origins and risk factors for SCD-related brain abnormalities. This will support development of preventive and supportive strategies as well as the initiation and evaluation of therapeutic interventions. Previous experience with the performance of brain MRI scans combined with recent research, indicates that the emotional burden placed on young children when undergoing a brain MR scan, are proportionate to the emotional burden placed on adults when they undergo a brain MR-scan. Furthermore, children will be offered the opportunity to become acquainted with the research procedure by witnessing an MRI scan session prior before participation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with SCD of all genotype between 6 and 18 at baseline

Exclusion Criteria:

* Parents/ guardians (in case of minors) or patients themselves (>16 years) unable to make an informed decision on participating in this study.

  * An abnormal brain MRI prior to initiation of the study due to non-SCD related causes.
  * Contraindications for brain MRI per protocol

Ages: 6 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents diagnosed with SCD of all genotypes, treated at Erasmus MC and the Amsterdam UMC, ranging from 6 to 18 years at initiation of the study.
  The clinical phenotype of SCD consists of a spectrum: From the patients with a high hemoglobin plus an absent or lower incidence of VOCs to the patients with a higher hemoglobin and a higher incidence of VOCs. We chose to include SCD patients of all genotypes, not only the HbSS and Hbẞ0 thalassemia, to cover the whole phenotypic range of SCD. This was chosen in order to infer the possible causes of an expected difference in white matter volume increase, like anemia and sickling-propensity.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
mm3/time unit | 4 years
  Total white matter volume increase in children and adolescents with SCD

SECONDARY OUTCOMES:
Full scale IQ (FSIQ) | 4 years
  Neurocognitive functioning (intelligence, specific neurocognitive functions, network organization)
Incidence of stroke | 4 years
Other forms complications due to SCD | 4 years
Amount of hospital admissions | 4 years
Ld, bilirubin | 4 years
  Hemolysis biomarkers
Times/year | 4 years
  ER visits
Hb, Ht | 4 years
  Biomarkers for anemia
T score metric: a score of 50 represents the mean score of a reference population and 10 is the standard deviation. | 4 years
  Patient-Reported Outcomes Measurement Information System® (PROMIS) within domains such as fatigue, pain behavior, depression, anxiety

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Erasmus MC, Rotterdam, South Holland
  - Amsterdam University Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: Undecided